CLINICAL TRIAL: NCT04389840
Title: A Phase 2/3 Study to Evaluate the Safety and Efficacy of Dociparstat Sodium for the Treatment of Severe COVID-19 in Adults at High Risk of Respiratory Failure
Brief Title: Dociparstat for the Treatment of Severe COVID-19 in Adults at High Risk of Respiratory Failure
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to improvement in the Coronavirus Disease 2019 (COVID-19) pandemic and low subject accrual.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMX-DS-004
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Coronavirus Disease 2019 (COVID-19); Acute Lung Injury; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Keywords: COVID-19; ALI; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Acute Lung Injury | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The first 12 subjects were to be randomized 1:1 (dociparstat:placebo) All other subjects were to be randomized 2:1 (dociparstat:placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 dociparstat (Experimental): Subjects received 4 mg/kg of dociparstat administered as an intravenous (IV) bolus on Day 1, followed by 0.25 mg/kg/hr dociparstat by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
  Interventions: Drug: Dociparstat sodium
- Cohort 1 placebo (Placebo Comparator): Placebo IV bolus on Day 1, followed by Placebo by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours])
  Interventions: Drug: Placebo
- Cohort 2 dociparstat (Experimental): Subjects received 4 mg/kg of dociparstat administered as an intravenous (IV) bolus on Day 1, followed by 0.325 mg/kg/hr dociparstat by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
  Interventions: Drug: Dociparstat sodium
- Cohort 2 placebo (Placebo Comparator): Subjects received placebo IV bolus on Day 1, followed by placebo by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
  Interventions: Drug: Placebo
- Cohort 3 dociparstat (Experimental): Subjects received 4 mg/kg of dociparstat administered as an intravenous (IV) bolus on Day 1, followed by 0.325 mg/kg/hr dociparstat by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
  Interventions: Drug: Dociparstat sodium
- Cohort 3 placebo (Placebo Comparator): Subjects received placebo IV bolus on Day 1, followed by placebo by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dociparstat sodium — Dociparstat is a glycosaminoglycan derived from porcine heparin.
  Other Names: DSTAT; CX-01; 2-0,3-0 desulfated heparin; ODSH
  Arms: Cohort 1 dociparstat; Cohort 2 dociparstat; Cohort 3 dociparstat
Drug: Placebo — 0.9% Normal Saline
  Other Names: Normal saline; Sodium chloride 0.9%; 0.9% Normal Saline
  Arms: Cohort 1 placebo; Cohort 2 placebo; Cohort 3 placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled Phase 2/3 study to evaluate the safety and efficacy of dociparstat sodium in adult patients with acute lung injury (ALI) due to Coronavirus Disease 2019 (COVID-19). This study was designed to determine if dociparstat sodium could accelerate recovery and prevent progression to mechanical ventilation in patients severely affected by COVID-19.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, Phase 2/3 trial to evaluate the safety and efficacy of dociparsat sodium in adults patients with severe COVID-19 who were at high risk of respiratory failure. Eligible subjects were with confirmed COVID-19 and required hospitalization and supplemental oxygen therapy. This study was designed to determine if dociparstat sodium could accelerate recovery and prevent progression to mechanical ventilation in patients severely affected by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

A potential participant must have met all the following criteria to be included in the study:

1. Was hospitalized for laboratory-documented Coronavirus Disease 2019 (COVID-19) (e.g., positive for severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] via nasopharyngeal swab real time polymerase chain reaction [RT-PCR; or other commercial or public health assay]).
2. Was aged ≥18 years and ≤85 years.
3. Had a resting oxygen saturation (SaO2) of <94% while breathing ambient air.
4. Had a score of 3 or 4 on the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale (required supplemental oxygen or non-invasive ventilation).
5. Had provided informed consent to participate in the study (by participant or legally-acceptable representative).

Exclusion Criteria:

A potential participant who met any of the following criteria was not eligible to participate in the study:

1. Was currently receiving invasive mechanical ventilation (e.g., via an endotracheal tube) (score of 2 on NIAID ordinal scale).
2. Had severe chronic respiratory disease, defined by any oxygen requirement prior to incident COVID-19.
3. Had active or uncontrolled bleeding at the time of randomization; a bleeding disorder, either inherited or caused by disease; history of known arterial-venous malformation, intracranial hemorrhage, or suspected or known cerebral aneurysm; or clinically significant (in the judgment of the Investigator) gastrointestinal bleeding within the 3 weeks prior to randomization.
4. Was receiving any other investigational (non-approved) therapy for the treatment of COVID-19 or participating in the treatment period of any other therapeutic intervention clinical study. Participating in the follow-up period of an interventional study may be permitted with prior medical monitor approval; participation in an observational study is permitted.
5. Was receiving systemic corticosteroids for a chronic condition.
6. Was receiving chronic anticoagulation with warfarin or direct oral anticoagulants (e.g., rivaroxaban, dabigatran, apixaban, edoxaban).
7. Was receiving or anticipated to require other systemic anticoagulation dosing at a therapeutic intensity. Prophylaxis of venous thromboembolism (VTE) using subcutaneous (SC) unfractionated heparin or enoxaparin was permitted with appropriate monitoring of coagulation status and within the guidelines described in the protocol.
8. Was receiving antiplatelet therapy, alone or in combination, including aspirin and other antiplatelet agents (e.g., clopidogrel, ticagrelor, and prasugrel), unless able to discontinue these agents at the time of randomization and was able to remain off these agents throughout the duration of the study intervention infusion period.
9. Had treatment with systemic (non-steroid) immunomodulators or immunosuppressant medications, including but not limited to tumor necrosis factor (TNF) inhibitors, anti-interleukin-1 agents and Janus kinase (JAK) inhibitors within 5 half-lives or 30 days (whichever was longer) prior to randomization.
10. Had a history of congestive heart failure requiring hospitalization.
11. Had active pericarditis (based on clinical assessment).
12. Had malignancy or other irreversible disease or condition for which 6-month mortality was estimated ≥50%.
13. Had a corrected QT interval (QTc) >500 msec (or >530-550 msec in participants with QRS greater than >120 msec).
14. Had a Tisdale risk score ≥11 without the ability to monitor with serial electrocardiograms (ECGs) or telemetry.
15. Had severe renal impairment, as determined by calculated creatinine clearance <30 mL/min or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2.
16. Had alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >5x upper limit of normal (ULN).
17. Had activated partial thromboplastin time (aPTT) >42 seconds.
18. Had thrombocytopenia with a platelet count <80,000/mm3.
19. Had severe chronic liver disease (Child-Pugh Score of 10 to 15).
20. Had received dociparstat in a different clinical study.
21. Woman of childbearing potential who was pregnant, breastfeeding, and/or not using a highly-effective method of contraception (consistent with local regulations regarding the methods of contraception for those participating in clinical studies).
22. Had evidence of clinical improvement in COVID-19 status including, but not limited to, a sustained reduction in oxygen requirements over the previous 48 hours, or extubated and/or no longer requiring mechanical ventilation following intubation for COVID-19.
23. Had any other condition, including abnormal laboratory values, that, in the judgment of the Investigator, could have put the participant at increased risk, or would have interfered with the conduct or planned analysis of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Advanced Pulmonary Research Institute/Wellington Regional Medical Center, Loxahatchee Groves, Florida
  - Augusta University, Augusta, Georgia
  - Our Lady of the Lake, Baton Rouge, Louisiana
  - Tulane University, New Orleans, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - Ascension Macomb-Oakland Cardiovascular Research, Warren, Michigan
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Texas Health Harris Methodist Hospital Fort Worth, Dallas, Texas
  - Ascension St. Francis Hospital, Milwaukee, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasky JA, Fuloria J, Morrison ME, Lanier R, Naderer O, Brundage T, Melemed A. Design and Rationale of a Randomized, Double-Blind, Placebo-Controlled, Phase 2/3 Study Evaluating Dociparstat in Acute Lung Injury Associated with Severe COVID-19. Adv Ther. 2021 Jan;38(1):782-791. doi: 10.1007/s12325-020-01539-z. Epub 2020 Oct 27. PMID 33108622
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrollment was terminated on 20 May 2021 due to improvement in the Coronavirus Disease 2019 (COVID-19) pandemic and low subject accrual. At the time of termination, a total of 27 subjects of the planned 75 subjects had been enrolled, of which 26 subjects were treated and 22 subjects had completed the study across Cohorts 1, 2, and 3 (partial) of the Phase 2 portion of the study.
Groups:
- Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 Placebo: Subjects received placebo IV bolus on Day 1, followed by placebo by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
Period: Overall Study
Arm/Group | Cohort 1 Dociparstat | Cohort 1 Placebo | Cohort 2 Dociparstat | Cohort 2 Placebo | Cohort 3 Dociparstat | Cohort 3 Placebo
Started | 6 | 6 | 8 | 4 | 2 | 1
Intent-to-Treat Analysis Set | 6 | 6 | 8 | 4 | 2 | 1
Safety Analysis Set | 6 | 6 | 8 | 3 (The excluded subject was randomized to receive placebo but never received treatment due to consent withdrawal.) | 2 | 1
Completed | 4 | 5 | 8 | 3 | 1 | 1
Not Completed | 2 | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject request and prohibited concomitant medication | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Note: Baseline characteristics were evaluated for the Safety Analysis Set. The Intent-to-Treat Analysis Set included 4 placebo-treated subjects from Cohort 2; however, only 3 placebo-treated subjects from Cohort 2 were included in the Safety Analysis Set. The excluded subject was randomized to receive placebo but never received treatment due to consent withdrawal.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Dociparstat | Cohort 1 Placebo | Cohort 2 Dociparstat | Cohort 2 Placebo | Cohort 3 Dociparstat | Cohort 3 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 8 | 3 | 2 | 1 | 26
Age, Continuous [Median (Full Range); unit: years] | 50.5 [32 to 67] | 63.0 [47 to 70] | 62.0 [36 to 66] | 62.0 [56 to 65] | 39.5 [38 to 41] | 41 [41 to 41] | 57.0 [32 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 3 | 0 | 0 | 15
  Male | 0 | 2 | 6 | 0 | 2 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 0 | 1 | 9
  White | 4 | 4 | 4 | 1 | 1 | 0 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 0 | 2
NIAID Score (actual) [Count of Participants; unit: Participants] — NIAID Score (actual) was calculated using hospitalization and ventilation status at the time of randomization. The ordinal scale is an assessment of the clinical status of the participant at a given time point. Scores 3 and 4 are as follows:
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices. 4. Hospitalized, requiring supplemental oxygen.
  Participants
    3 | 2 | 5 | 2 | 0 | 2 | 1 | 12
    4 | 4 | 1 | 6 | 3 | 0 | 0 | 14
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (6.57) | 33.9 (5.85) | 31.0 (6.17) | 36.4 (12.34) | 28.6 (5.05) | 45.4 (NA) — There was only 1 subject in this cohort. | 33.0 (6.85)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Alive and Free of Invasive Mechanical Ventilation or ECMO Through Day 28
Description: The primary efficacy endpoint was to be the proportion of participants who were alive and free of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) through Day 28. Data also shows proportion of participants with invasive mechanical ventilation or ECMO, all-cause mortality, or early study discontinuation (<Day 25), whichever occurred first, by Day 28.
Time Frame: Day 1 to Day 28 (28 days)
Population: Note: This outcome measure was analyzed using the Intent-to-Treat (ITT) Analysis Set. In the ITT Analysis Set included 4 placebo-treated subjects for Cohort 2; however, only 3 placebo-treated subjects from Cohort 2 were included in the Safety Analysis Set. This subject was randomized to receive placebo but never received treatment due to consent withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Dociparstat | Cohort 1 Placebo | Cohort 2 Dociparstat | Cohort 2 Placebo | Cohort 3 Dociparstat | Cohort 3 Placebo
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 2 | 1
Participants | 3 | 4 | 7 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: From randomization through Day 28
Description: Note: Adverse events were evaluated using the Safety Analysis Set. All-cause mortality was evaluated using the Intent-to-Treat (ITT) Analysis Set. The ITT Analysis Set included 4 placebo-treated subjects from Cohort 2; however, only 3 placebo-treated subjects from Cohort 2 were included in the Safety Analysis Set. The excluded subject was randomized to receive placebo but never received treatment due to consent withdrawal.
Groups:
- Cohort 3 Placebo: Subjects received 4 mg/kg of dociparstat administered as an intravenous (IV) bolus on Day 1, followed by 0.325 mg/kg/hr dociparstat by continuous IV infusion for 24 hours daily for up to 7 days (starting on Day 1 and ending on Day 8 [168 hours]).
Arm/Group | Cohort 1 Dociparstat | Cohort 1 Placebo | Cohort 2 Dociparstat | Cohort 2 Placebo | Cohort 3 Dociparstat | Cohort 3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 0/8 | 0/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 1/8 | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/8 | 2/3 | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Dociparstat (N=6) | Cohort 1 Placebo (N=6) | Cohort 2 Dociparstat (N=8) | Cohort 2 Placebo (N=3) | Cohort 3 Dociparstat (N=2) | Cohort 3 Placebo (N=1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Dociparstat (N=6) | Cohort 1 Placebo (N=6) | Cohort 2 Dociparstat (N=8) | Cohort 2 Placebo (N=3) | Cohort 3 Dociparstat (N=2) | Cohort 3 Placebo (N=1)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorous decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to improvement in the Coronavirus Disease 2019 (COVID-19) pandemic and low subject accrual, study enrollment was prematurely terminated on 20 May 2021. Therefore, formal statistical analyses were not performed, and no conclusions can be drawn about docipartstat with regards to efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT04389840/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04389840/SAP_001.pdf